CLINICAL TRIAL: NCT00204906
Title: Effect of Vitamin D Supplementation on Skeletal and Overall Health of Nursing Home Residents
Brief Title: Correction of Vitamin D Inadequacy in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2004-0057
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-06

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency

INTERVENTIONS:
Dietary Supplement: vitamin D supplementation

SUMMARY:
Vitamin D inadequacy continues to be neglected in nursing home residents. We hypothesized that part of this neglect is due to absence of data documenting safe and effective ways to replete this inadequacy.

DETAILED DESCRIPTION:
Vitamin D inadequacy continues to be neglected in nursing home residents. We hypothesized that part of this neglect is due to absence of data documenting safe and effective ways to replete this inadequacy. Subjects with low vitamin D concentrations are dosed with 50.000 IU three times a week for 25 hydroxy vitamin D, parathyroid hormone and bone turnover status. .

ELIGIBILITY:
Inclusion Criteria:

* Able to walk
* Reside in nursing home for the 12 weeks of study

Exclusion Criteria:

* Non-ambulatory residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States